CLINICAL TRIAL: NCT02908451
Title: A Phase I Dose Escalation Study, With Cohort Expansion, to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AbGn-107 Therapy in Patients With Chemo-refractory Locally Advanced, Recurrent, or Metastatic Gastric, Colorectal, Pancreatic or Biliary Cancer
Brief Title: A Study of AbGn-107 in Patients With Gastric, Colorectal, Pancreatic or Biliary Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 pandemic has caused a huge operational difficulty for this ongoing clinical trial, as many hospitals have set limitations on onsite staff, patient visits, study related procedures and onsite monitoring visits.
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016.006.01
Record Dates: First submitted 2016-09-06; First posted 2016-09-21 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2020-07

CONDITIONS: Gastric Cancer; Colorectal Cancer; Pancreatic Cancer; Biliary Cancer
Keywords: Cancer; Antibody Drug Conjugate; AbGn-107; Adenocarcinoma; Gastric; Colorectal; Pancreatic; biliary; cholangiocarcinoma; gallbladder; ampullary carcinomas
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Neoplasms; Adenocarcinoma; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AbGn-107 (Experimental): AbGn-107 will be administered every 14-days or 28-days via intravenous infusion. Patients with a complete response (CR), partial response (PR), or stable disease (SD), or with evidence of clinical benefit may be treated every continuously every 14-days or 28-days..
  Interventions: Biological: AbGn-107

INTERVENTIONS:
Biological: AbGn-107 — Antibody Drug Conjugate

SUMMARY:
This study is to define the safety profile and to determine the Maximal tolerated dose regimen and preliminary efficacy of AbGn-107 administered every 14 days (Q2W regimen) or 28 days (Q4W regimen) in patients with chemo-refractory locally advanced, recurrent or metastatic gastric, colorectal, pancreatic or biliary cancer.

DETAILED DESCRIPTION:
AbGn-107 is an antibody drug conjugate (ADC) which targets an antigen (AG7 antigen) present in gastric, colorectal, pancreatic cancer or biliary cancer. This study is a standard 3 + 3 dose escalation design with cohort expansion. AbGn-107 will be administered every 14 days (Q2W regimen) or 28 days (Q4W regimen) in patients with chemo-refractory locally advanced, recurrent or metastatic gastric, colorectal, pancreatic adenocarcinoma or biliary cancer. The primary objectives of this study are to define the safety profile and to determine the maximum tolerated dose regimen of AbGn-107, and the secondary objectives are to evaluate the pharmacokinetic (PK) parameters, the immunogenicity, and preliminary efficacy of AbGn-107.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years. A patient may be of either sex and of any race/ethnicity.
2. Histologically confirmed, chemo-refractory, locally advanced, recurrent or metastatic gastric (including GE junction), colorectal, or pancreatic adenocarcinoma or biliary cancer (including cholangiocarcinoma, gallbladder and ampullary carcinomas).

   1. Patient must not have curative options available (e.g. a single metastatic focus in the liver in a patient with MCRC eligible for metastasectomy).
   2. Chemo-refractory is defined as:

      * Progression on or following, or intolerant of, at least one prior line of standard systemic therapy for advanced or metastatic gastric or pancreatic or biliary cancers.
      * Progression on or following, or intolerant of, at least two prior lines of standard systemic therapy for advanced or metastatic colorectal cancers.
      * Patients who have progressed/recurred following neoadjuvant/adjuvant chemotherapy for earlier stage disease, if completed within the previous 6 months, are eligible.
3. Archived tissue must be available for all patients (both dose escalation and expansion cohorts). Dose Escalation Only-If tissue is not available, patients may still be considered eligible for enrollment, if all other eligibility criteria are confirmed and after discussion with and approval by the sponsor medical monitor. Cohort Expansion Only-Tissue must be to confirmed high expression of AG7 antigen during the Pre-Screening period, defined as immune reactive score (IRS) ≥8, via slides from original diagnostic biopsy material or biopsy of recurrent/metastatic disease, prior to enrollment.
4. Measurable disease by RECIST 1.1 criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
6. Adequate organ function within 3 weeks prior to first study drug administration as evidenced by:

   1. Absolute neutrophil count ≥1.5 x 10^9/L,
   2. Hemoglobin ≥9 g/dL,
   3. Platelet count ≥100 x 10^9/L,
   4. Serum creatinine ≤1.5 x upper limit of normal (ULN) or a calculated creatinine clearance >60 mL/min,
   5. Total bilirubin <1.5 x ULN, except for patients with Gilbert's disease who are eligible if total bilirubin ≤ 3 mg/dL.
   6. Aspartate aminotransferase (AST)/serum glutamic-oxalacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <2.5 x ULN, or, in the presence of documented liver metastases, ≤5 x ULN.
7. Ability to adhere to dose and visit schedules.
8. Women of childbearing potential (WOCP) must have a negative pregnancy test result prior to enrollment. WOCP and men whose partners are WOCP must agree to use a highly effective method of birth control during the study and for 6 months following the last dose of study drug. A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).
9. Ability to provide written informed consent
10. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Any persistent, unresolved Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 drug-related toxicity (except alopecia, erectile impotence, tinnitus, hot flashes, and loss of libido) associated with previous treatment. Inclusion of patients with persistent neuropathy or hearing loss Grade ≥2 due to previous treatment requires discussion with the sponsor.
2. Radiation therapy within 2 weeks prior to first study drug administration.
3. Major surgery within 3 weeks prior to first study drug administration.
4. Any chemotherapy within 30 days of enrollment.
5. Participation in any other clinical study with a potentially therapeutic agent or receipt of another investigational product within 21 days or 5 plasma half-lives, whichever is longer, prior to first day of drug administration (Day 1).
6. Active central nervous system metastases. Patients with a history of brain metastases may be eligible, provided they have been definitively treated and are clinically stable, after discussion with sponsor. Treated or untreated leptomeningeal disease is not permitted.
7. Known human immunodeficiency virus (HIV) infection or a known HIV-related malignancy. Note: HIV testing is not required unless there is any clinical suspicion that the patient might be HIV positive.
8. Known active hepatitis B or C. HBV and HCV tests are required prior to Day 1.
9. Any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would impair with their ability to receive or tolerate the planned treatment, or interfere with the study evaluations or optimal participation in the study.
10. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) graded according to CTCAE v4.03. | 28 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | 70 days after treatment
Tmax (time from dosing to maximum measured concentration) | 70 days after treatment
T1/2 (half-life of the analyte) | 70 days after treatment
Immunogenicity evaluation based on anti-drug antibodies titer | 70 days after treatment
Overall Response Rate Evaluated by Response Evaluation Criteria in Solid Tumor (RECIST) | Every 2 treatment cycles for Q4W regimen or every 4 treatment cycles for Q2W regimen, up to 2 years from the first patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao (David) Lin, MD, PhD, Study Director — AbGenomics B.V.; Andrew Ko, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - University of California, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko AH, Coveler AL, Schlechter BL, Bekaii-Saab T, Wolpin BM, Clark JW, Bockorny B, Bai LY, Lin YC, Chiang E, Langecker P, Lin SY. A multicenter phase Ia study of AbGn-107, a novel antibody-drug conjugate, in patients with advanced gastrointestinal cancer. Invest New Drugs. 2024 Apr;42(2):221-228. doi: 10.1007/s10637-024-01430-6. Epub 2024 Mar 5. PMID 38441850